CLINICAL TRIAL: NCT06952478
Title: A Double-Blind, Randomized, Active-Controlled, Parallel-group, Phase 1/3 Study to Compare Pharmacokinetics, Efficacy and Safety of Subcutaneous CT-P44 and Darzalex Faspro in Combination With Lenalidomide and Dexamethasone in Patients With Refractory or Relapsed Multiple Myeloma
Brief Title: A Study to Compare Pharmacokinetics, Efficacy and Safety of Subcutaneous CT-P44 and Darzalex Faspro in Combination With Lenalidomide and Dexamethasone in Patients With Refractory or Relapsed Multiple Myeloma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P44 3.1; 2024-518588-36-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-29; First posted 2025-05-01 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Refractory or Relapsed Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CT-P44 (Experimental): CT-P44 1800mg SC (subcutaneous)
  Interventions: Biological: CT-P44(Daratumumab)
- Darzalex Faspro (Active Comparator): Darzalex Faspro 1800mg SC (subcutaneous)
  Interventions: Biological: Darzalex Faspro(Daratumumab)

INTERVENTIONS:
Biological: CT-P44(Daratumumab) — CT-P44 1800 mg will be administered as SC injection in combination with Rd until each patient's PD, unacceptable toxicity or Cycle 26, whichever occurs first.
  Arms: CT-P44
Biological: Darzalex Faspro(Daratumumab) — Darzalex Faspro 1800 mg will be administered as SC injection in combination with Rd until each patient's PD, unacceptable toxicity or Cycle 13, whichever occurs first.
  Arms: Darzalex Faspro

SUMMARY:
This study is a phase 1/3 study to Compare Pharmacokinetics, Efficacy and Safety of Subcutaneous CT-P44 and Darzalex Faspro in Combination with Lenalidomide and Dexamethasone in Patients with Refractory or Relapsed Multiple Myeloma

ELIGIBILITY:
[Main Inclusion Criteria]

* Male or female with 18 years of age or older.
* Patient must have documented multiple myeloma (MM) according to IMWG criteria
* Patient must have a documented relapsed or refractory disease.
* Patient must have achieved a response (PR or better based on investigator's determination of response by the IMWG criteria) to at least one prior regimen.
* Patient must have a PD as defined by the IMWG criteria on or after their last line of therapy.

[Main Exclusion Criteria]

* Patient has received daratumumab or any other drug specifically targeting CD38 previously.
* Patient's disease shows evidence of refractoriness or intolerance to lenalidomide.
* Patient is known or suspected of not being able to comply with the study protocol (e.g., psychological disorder) or the patient has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the patient (e.g., compromise their well-being) or that could prevent, limit, or confound the protocol-specified assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2029-06-25 (Estimated)

PRIMARY OUTCOMES:
PK equivalence of CT-P44 and Darzalex Faspro | Week 0 ~ Week 24
  AUCWeek0-1 and AUCWeek8-10 of daratumumab.
Therapeutic equivalence of CT-P44 and Darzalex Faspro | Week 0 ~ Week 24
  Proportion of patients who will achieve VGPR or better (sCR + CR + VGPR) based on the confirmed BOR.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Beitou District, Taiwan